CLINICAL TRIAL: NCT02672904
Title: Comparison Between the Use of KTP Laser vs. CO2 Laser for Endoscopic Surgical Removal of Malignant Neoplasms of the Vocal Cords
Brief Title: KTP vs CO2 Laser for the Treatment of Laryngeal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Dr Yonatan Lahav, Dr Yonatan Lahav, Kaplan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0057-11-KMC-CTIL
Record Dates: First submitted 2016-01-26; First posted 2016-02-03 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Laryngeal Neoplasms
Keywords: vocal cord; carcinoma; ktp laser; co2 laser; endoscopic surgery
MeSH Terms: conditions — Laryngeal Neoplasms; Carcinoma | interventions — Lasers, Gas; Lasers, Solid-State

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CO2 laser (Active Comparator): Patients undergoing endoscopic treatment with CO2 laser
  Interventions: Device: CO2 laser
- KTP laser (Active Comparator): Patients undergoing endoscopic treatment with KTP laser
  Interventions: Device: KTP laser

INTERVENTIONS:
Device: CO2 laser — surgical removal of carcinoma from the vocal cords with CO2 laser
  Arms: CO2 laser
Device: KTP laser — surgical removal of carcinoma from the vocal cords with KTP laser
  Arms: KTP laser

SUMMARY:
comparison results of treatment of early stage glottic cancer between two methods of surgical treatment - CO2 laser and KTP laser

DETAILED DESCRIPTION:
Randomized controlled double-blinded study. The study group includes patients diagnosed with early glottic cancer, either carcinoma in situ or T1a-b,N0M0 squamous cell carcinoma.

Patients will undergo examination and treatment and at least 3 years of follow-up.

40 cancer patients will be included. The participants will be randomly divided into two groups: the first will be treated by KTP laser and the second by CO2 laser.

The patients will be blinded to the method of treatment. To enable double-blinding, the investigator performing the surgery would be the only one knowing which research group the patient belongs to. The investigator in charge of collecting the data after the operation will be blinded to the treatment method.

Each participant will undergo pre-operative evaluation and follow-up after surgery in both arms.

Preoperative evaluation will include:

* Voice Handicap Index questionnaire
* GRBAS - subjective assessment of voice quality.
* Video-stroboscopy of vocal cords
* Voice Analysis .

Follow-up after surgery:

* Visit 6 weeks after surgery (± two weeks), and then every three months (± 6 weeks).
* repeated full evaluation (questionnaire, GRBAS, Stroboscopy, voice analysis) in 30 weeks of follow up and 3 years of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pre-operative diagnosis of squamous cell cancer of the vocal cords at an early stage ( Carcinoma in situ or T1-glottic carcinoma).

Exclusion Criteria:

* Patients who underwent previous significant vocal cords surgical intervention , or irradiation.
* Contraindications to any endoscopic surgical treatment (general health condition, patient refusal, technical surgical difficulties)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Duration of surgery | intraoperative
  total time (minutes) of surgical procedure
number of surgical interventions | 3 years
  total number of surgical interventions needed to eliminate the disease
Recovery time after surgery | up to 3 years
  recovery in terms of overall function, breathing, swallowing and vocal communication
voice quality results In the short term | 6 month after last intervention
  objective measurement- voice lab analysis, and subjective measurement- Voice Handicap Index questionnaire
voice quality results In the long term | 3 years after last intervention
  objective measurement- voice lab analysis, and subjective measurement- Voice Handicap Index questionnaire
Cure rates in terms of local, regional or distant recurrence events | 3 years after last intervention
  evidence of malignant disease in the larynx, cervical lymph nodes or distant metastases
Overall survival and disease-dependent survival over a period of at least 3 years | 3 years after last intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yonatan Lahav, Dr, Principal Investigator — Kaplan Medical Center
Locations (1):
- Kapkan medical center, Rehovot, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burns JA, Friedman AD, Lutch MJ, Hillman RE, Zeitels SM. Value and utility of 532 nanometre pulsed potassium-titanyl-phosphate laser in endoscopic laryngeal surgery. J Laryngol Otol. 2010 Apr;124(4):407-11. doi: 10.1017/S0022215109991824. Epub 2009 Nov 27. PMID 19941682
- [Background] Zeitels SM, Burns JA, Lopez-Guerra G, Anderson RR, Hillman RE. Photoangiolytic laser treatment of early glottic cancer: a new management strategy. Ann Otol Rhinol Laryngol Suppl. 2008 Jul;199:3-24. doi: 10.1177/00034894081170s701. PMID 18710131
- [Background] Lin DS, Cheng SC, Su WF. Potassium titanyl phosphate laser treatment of intubation vocal granuloma. Eur Arch Otorhinolaryngol. 2008 Oct;265(10):1233-8. doi: 10.1007/s00405-008-0628-6. Epub 2008 Mar 4. PMID 18317789
- [Background] Zeitels SM, Akst LM, Bums JA, Hillman RE, Broadhurst MS, Anderson RR. Pulsed angiolytic laser treatment of ectasias and varices in singers. Ann Otol Rhinol Laryngol. 2006 Aug;115(8):571-80. doi: 10.1177/000348940611500802. PMID 16944655
- [Background] Hirano S, Yamashita M, Kitamura M, Takagita S. Photocoagulation of microvascular and hemorrhagic lesions of the vocal fold with the KTP laser. Ann Otol Rhinol Laryngol. 2006 Apr;115(4):253-9. doi: 10.1177/000348940611500402. PMID 16676821
- [Background] Kacker A, April M, Ward RF. Use of potassium titanyl phosphate (KTP) laser in management of subglottic hemangiomas. Int J Pediatr Otorhinolaryngol. 2001 May 31;59(1):15-21. doi: 10.1016/s0165-5876(01)00451-7. PMID 11376814
- [Background] Zeitels SM, Burns JA. Office-based laryngeal laser surgery with the 532-nm pulsed-potassium-titanyl-phosphate laser. Curr Opin Otolaryngol Head Neck Surg. 2007 Dec;15(6):394-400. doi: 10.1097/MOO.0b013e3282f1fbb2. PMID 17986877
- [Background] Zeitels SM, Akst LM, Burns JA, Hillman RE, Broadhurst MS, Anderson RR. Office-based 532-nm pulsed KTP laser treatment of glottal papillomatosis and dysplasia. Ann Otol Rhinol Laryngol. 2006 Sep;115(9):679-85. doi: 10.1177/000348940611500905. PMID 17044539